CLINICAL TRIAL: NCT06170879
Title: What is the Experience of the Professional Nurse Advocates (PNAs) Application of the A-EQUIP Model Into Practice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: LPR 3286
Record Dates: First submitted 2023-12-01; First posted 2023-12-14 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-05

CONDITIONS: Staff Attitude; Professional Role

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will utilise focus groups with trained PNAs from different Trusts spread over the Midlands region within England. This approach will help explore the experiences and views of trained PNAs in the application of the role and the foundations on which it is supported. It will also supply valuable feedback regarding the preparation, implementation, and outcome of adopting the PNA position with health care organisations, as there is a suggestion that the role could expand from England to the United Kingdom and possibly the United States of America.

ELIGIBILITY:
Inclusion Criteria:

• Qualified Professional Nurse Advocate (PNAs) all of whom would have successfully completed a PNA level 7 module provided by a Higher Education Institution within England

Exclusion Criteria:

• Any qualified nurse who has not successfully completed a PNA module.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Professional nurse advocates working in the Midlands
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
To measure the experiences of PNAs in implementing the role within their clinical practice and using the A-EQUIP model | 3 months
  To explore the experiences of Professional Nurse Advocates and their application of the A-EQUIP model into clinical practice

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, United Kingdom